CLINICAL TRIAL: NCT04861428
Title: Initial Cross-over Test of a Heat-not-burn Tobacco Product to Aid in Switching From Combustible to Noncombustible Nicotine in Smokers
Brief Title: Heat-not-burn Tobacco Product to Aid in Switching From Combustible to Noncombustible Nicotine (IQOS)
Acronym: IQOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution and did not retain the study
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jian-Min Yuan, MD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HCC 20-245
Record Dates: First submitted 2021-04-13; First posted 2021-04-27 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Smoking Behaviors
Keywords: HnB: heat not burn tobacco product; IQOS: commercially available HnB manufactured
MeSH Terms: conditions — Smoking | interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQOS / Smoking as usual (Experimental): Two weeks of IQOS, followed by two weeks of cigarette smoking as usual.
  Interventions: Other: IQOS; Other: Smoking as Usual
- Smoking as usual / IQOS (Active Comparator): Two weeks of cigarette smoking as usual, followed by two weeks of IQOS.
  Interventions: Other: IQOS; Other: Smoking as Usual

INTERVENTIONS:
Other: IQOS — IQOS is a heat-not-burn tobacco product (consisting of an electronic heating device and Heatstick tobacco rods).
Other: Smoking as Usual — Cigarette smoking

SUMMARY:
A novel heat-not-burn tobacco product (IQOS) will be provided to smokers, compared against a (cigarette) smoking as usual period in counter-balanced order in a cross-over design. This study will examine the short-term effects of IQOS, switching from combustible to noncombustible nicotine and withdrawal-related symptoms over a two week-long "practice" period, relative to smoking as usual.

DETAILED DESCRIPTION:
The current within-subjects crossover study aims to directly compare initial efficacy of IQOS vs (cigarette) smoking as usual on switching from tobacco cigarettes during two-week "practice" periods in smokers.

Study interventions include IQOS, a commercially available, over the counter product. The IQOS is a commercially available tobacco product that consists of a holder which contains a rechargeable battery and an electronically heated metal blade.

All procedures will take place in the Prevention and Early Detection Center (PEDC) at the UPMC Hillman Cancer Center. Participants will be assessed daily via remote CO assessment and online questionnaire throughout the entire study (WK1-WK5). At the end of a one-week baseline of normal smoking (WK1), participants will be randomized to either: 1) begin a two-week period of attempting to completely switch to exclusive IQOS use (IQOS First); or 2) continue to smoke as usual (IQOS Last; WK2-WK3), followed by a second two-week period during which they will smoke as usual or attempt to switch to IQOS (opposite of the first period; WK4-WK5).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 21-77
* Current smoker with ≥5 cigarettes per day for ≥1 year history of smoking
* Screening CO ≥8 ppm
* Not currently interested in quitting smoking
* Willing to briefly switch from combustible to noncombustible nicotine
* Have reliable daily access to a smartphone or tablet compatible with the iCO Smokerlyzer app:

  * Android 8 or higher, iOS 8 or higher
  * Bluetooth-enabled device

Exclusion Criteria:

* Current use of smoking cessation medications such as varenicline or bupropion
* Major chronic medical problems, including cardiovascular disease, diabetes
* Pregnancy (a urine pregnancy test will be administered at screening for all women of child bearing potential).

Ages: 21 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Objective smoke exposure | Up to 5 weeks
  Assessed daily using a mobile carbon monoxide monitor (iCO) provided to participants. Carbon monoxide (CO) readings parts per million (ppm) will be submitted directly via email using the iCO smartphone app.
Self-reported smoke exposure | Up to 5 weeks
  Assessed daily using self-reported cigarette consumption, with values submitted via online Qualtrics survey.
Harm exposure - Lung function | Up to 5 weeks
  Lung function will be assessed using standard pulmonary function test.
Harm exposure - Blood pressure | Up to 5 weeks
  Blood pressure will be assessed using a sphygmomanometer.

SECONDARY OUTCOMES:
Cigarette craving | Up to 5 weeks
  Cigarette craving measured daily via Qualtrics using the Questionnaire of Smoking Urges Brief version. This will be measured on a 0-100 visual analog scale. Higher scored indicate greater craving.
Withdrawal symptoms | Up to 5 weeks
  Withdrawal symptoms measured daily via Qualtrics using the Minnesota Nicotine Withdrawal Scale. This will be measured on a 0-18 scale. Higher scores indicate greater withdrawal symptoms.

OTHER OUTCOMES:
Complete switching | Up to 2 weeks
  Determined by the proportion of days where combination of CO values <7 ppm and zero self-reported cigarettes per day during the IQOS period.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No